CLINICAL TRIAL: NCT05913037
Title: A Randomized, Double-Blind, Placebo-Controlled, Multi-center Phase III Clinical Study to Evaluate the Efficacy and Safety of FCN-159 in Adult Patients With Symptomatic, Inoperable Neurofibromatosis Type 1-Related Plexiform Neurofibromas
Brief Title: FCN-159 in Adult Patients With Symptomatic, Inoperable Neurofibromatosis Type 1-Related Plexiform Neurofibromas
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Fosun Pharmaceutical Industrial Development Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FCN-159-007
Record Dates: First submitted 2023-06-06; First posted 2023-06-22 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Neurofibromatosis 1; Plexiform Neurofibroma; NF1
MeSH Terms: conditions — Neurofibromatosis 1; Neurofibroma, Plexiform | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FCN-159 (Experimental): Experimental: FCN-159 Dosage form:tablet Specification: 1mg，4mg Dose: FCN-159 8 mg, orally, once daily Method of administration: Oral
  Interventions: Drug: Test group (Group A): FCN-159 8 mg, orally, once daily;
- placebo (Placebo Comparator): Experimental: placebo Dosage form:tablet Specification: 1mg，4mg Dose: placebo 8 mg, orally, once daily Method of administration: Oral
  Interventions: Drug: Control group (Group B): Placebo, orally, once daily;

INTERVENTIONS:
Drug: Test group (Group A): FCN-159 8 mg, orally, once daily; — After completing all screening visit items, qualified patients will be randomly assigned to the test group (Group A) or control group (Group B) in a 2:1 ratio, and receive FCN-159 or placebo within 3 days after randomization.
  Arms: FCN-159
Drug: Control group (Group B): Placebo, orally, once daily; — After completing all screening visit items, qualified patients will be randomly assigned to the test group (Group A) or control group (Group B) in a 2:1 ratio, and receive FCN-159 or placebo within 3 days after randomization.
  Arms: placebo

SUMMARY:
A study to evaluate the efficacy of FCN-159 in adult patients with symptomatic, inoperable neurofibromatosis type 1-related plexiform neurofibromas.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, multi-center phase III clinical study to evaluate the efficacy and safety of FCN-159 in adult patients with symptomatic, inoperable neurofibromatosis type 1-related plexiform neurofibromas.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old and ≤ 70 years old.
2. Patients must be diagnosed with symptomatic NF1-related plexiform neurofibromas (PNs) and require systemic therapy at the investigator's discretion.
3. Presence of measurable lesions, defined as ≥ 3 cm in length in at least one dimension, which can be evaluated for efficacy by MRI.
4. Karnofsky performance status score ≥ 70.
5. Patients with adequate organ and bone marrow functions.

Exclusion Criteria:

1. NF1-related malignancies requiring chemotherapy, radiotherapy, or surgery, such as medium to high grade optic glioma or malignant peripheral nerve sheath tumor.
2. Patients with a history of or concurrently with other malignancies (excluding cured non-melanoma skin basal cell carcinoma, breast cancer in situ or cervical cancer in situ, and other malignancies without evidence of disease within 5 years).
3. Patients who cannot undergo MRI and/or have contraindications to MRI.
4. Patients with previous or current retinal vein obstruction (RVO), retinal pigment epithelial detachment (RPED), glaucoma, and other abnormal ophthalmic examination with clinical significance.
5. Interstitial pneumonia, including clinically significant radiation pneumonia.
6. Cardiac function or combined diseases meet one of the following conditions:

   1. QTcF value of > 470 milliseconds; patients with risk factors for QTcF prolongation or patients receiving drugs that prolong the QTcF interval.
   2. Congestive heart failure per New York Heart Association (NYHA) classification ≥ Class 3.
   3. Arrhythmias with clinical significance.
   4. Known concurrent clinically significant coronary artery disease, cardiomyopathy, and severe valvular disease.
   5. LVEF < 50%.
   6. Patients with a heart rate of < 50 beats/min.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2025-08-19 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) evaluated by BIRC (Response evaluation in Nerufibromatosis and Schwannomatosis, REiNS criteria) | Through study completion, an average of 2 years
  ORR is defined as the proportion of patients who have a confirmed complete response or confirmed partial response as determined by ICR per REiNS criteria.

SECONDARY OUTCOMES:
Objective response rate (ORR) evaluated by the investigator (REiNS criteria) | Through study completion, an average of 2 years
  ORR is defined as the proportion of patients who have a confirmed complete response or confirmed partial response as determined by ICR per REiNS criteria.
Duration of response (DOR) evaluated by BIRC and the investigator; | Through study completion, an average of 2 years
  DOR is defined as the time from the date of first documented response (which is subsequently confirmed) until progression by BIRC and the investigator per REiNS criteria or death due to any cause.
Disease control rate (DCR) evaluated by BIRC and the investigator; | Through study completion, an average of 2 years
  DCR is defined as the proportion of patients who have a confirmed complete response or confirmed partial response or stable disease as determined by BIRC and the investigator per REiNS criteria.
Clinical benefit rate (CBR)evaluated by BIRC and the investigator; | Through study completion, an average of 2 years
  CBR is defined as the proportion of patients who have a confirmed complete response or confirmed partial response or stable disease>48 weeks as determined by BIRC and the investigator per REiNS criteria.
Progression free survival (PFS) evaluated by BIRC and the investigator; | Through study completion, an average of 2 years
  PFS is defined as the time from randomization until date of disease progression by BIRC and investigator per REiNS criteria or death due to any cause.
Time to progression (TTP) evaluated by BIRC and the investigator; | Through study completion, an average of 2 years
  TTP is defined as the time from randomization until date of disease progression by BIRC and investigator per REiNS criteria.
Time to response (TTR) evaluated by BIRC and the investigator; | Through study completion, an average of 2 years
  TTR is defined as the time from date of randomization until the date of objective response by BIRC and investigator per REiNS criteria.
Change from baseline in pain intensity score | Through study completion, an average of 2 years
  Difference in mean change from baseline in overall tumor and target PN pain intensity score between Arm A and Arm B as assessed by the 11-point Numerical Rating Scale (NRS-11),which uses the range 0-10,higher scores mean worse outcome.
Change from baseline in appearance | Through study completion, an average of 2 years
  Change in appearance from baseline for Arm A versus Arm B as assessed using a sponsor-customized 'appearance evaluation'PRO questionnaire, which is descriptive.

CONTACTS AND LOCATIONS:
Overall Officials: Wenbin Li, MD, Principal Investigator — Beijing Tiantan Hospital
Locations (15):
- China (15):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Chinese Academy of Medical Sciences & Peking Union Medical College, Beijing, Beijing Municipality
  - Plastic Surgery Hospital,Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - TongJi Hospital，TongJi Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - The First Hospial of China Medical University, Shenyang, Liaoning
  - Fudan University Shanghai Cancer center, Shanghai, Shanghai Municipality
  - West China Hospital，Sichuan University, Chengdu, Sichuan
  - Hangzhou First People's Hospital, Hangzhou, Zhejiang
  - Zhejiang Provincial People'S Hospital, Hanzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No